CLINICAL TRIAL: NCT02328859
Title: Virtual Reality for Rehabilitation for Individuals With Lower Limb Amputation
Brief Title: Virtual Reality Rehabilitation for Individuals With Lower Limb Amputation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1598-P
Record Dates: First submitted 2014-12-09; First posted 2014-12-31 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Transtibial Amputation
Keywords: Gait; Rehabilitation; Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality gait rehabilitation (Experimental): Subjects will be trained using a custom treadmill with a virtual environment
  Interventions: Other: Virtual Reality Gait Training
- Treadmill training gait rehabilitation (Active Comparator): Subjects wil be trained using a standard treadmill without any visual display
  Interventions: Other: Treadmill Gait Training

INTERVENTIONS:
Other: Virtual Reality Gait Training — A Virtual Gait Retraining System (VGRS) will be used to train amputees for six weeks. the system consists of an actuated treadmill, a virtual environment and an avatar
  Arms: Virtual reality gait rehabilitation
Other: Treadmill Gait Training — A conventional treadmill with no visual display will be used to gait train amputees for a period of six weeks.
  Arms: Treadmill training gait rehabilitation

SUMMARY:
A custom designed Virtual Gait Retraining System (VGRS) is being adapted for balance and mobility rehabilitation in individuals with transtibial amputation. The system is composed of a treadmill that can simulate different environmental situations such as walking up stairs and hills and going around curves. The treadmill is synchronized with an immersive display and an avatar of the user. The combination of variable terrain and visual feedback is extremely promising as a means for amputee patients to achieve improved functional mobility after gait training. The proposed work is relevant to public health because it is the first step in developing a novel rehabilitation system that will use visual feedback for gait training in amputees and others with pathological gait disorders. The research is pertinent to the mission of the Department of Veterans Affairs which is committed to improve the quality of life of Veterans with disability.

DETAILED DESCRIPTION:
Lower extremity amputation can cause impairments in gait and balance due to the loss of proprioception and motor control. The asymmetries present during amputee gait are thought to be one of the major contributors to secondary musculoskeletal problems such as osteoarthritis. After lower extremity amputation, physical rehabilitation is necessary to achieve functional ambulation; however, no an evidence-based standard of care exists for individuals who undergo transtibial (TT) amputations. The objective of this application is to determine the effectiveness of gait training in an immersive virtual environment in people with transtibial amputation. The investigators' custom designed Virtual Gait Retraining System (VGRS) is a virtual reality (VR) system which provides visual and motor challenges while treadmill walking. The VGRS immerses the user in a virtual world, provides additional feedback with an avatar and presents the user with challenging tasks such as inclines and stair climbing which are complemented by the movement of the treadmill. The central hypothesis is that people with amputations will achieve greater improvements in balance, mobility and gait function using the investigators' custom designed VGRS as compared to current conventional treadmill gait training. This objective will be accomplished by addressing the following specific aims:

* 1) Compare the efficacy of VGRS to conventional treadmill training.
* 2) Evaluate the rate of improvement over the course of each training program (VGRS and conventional treadmill).

The investigators will conduct a randomized clinical trial with twenty TT amputee subjects comparing 6 weeks of training with the VGRS to 6 weeks of training using a conventional treadmill protocol. The investigators will use gait analysis, postural sway and standard balance and mobility instruments including the 6-Minute Walk Test, Four Square Step Test, the Berg Balance Scale and the Dynamic Gait Index to assess improvements in gait and mobility. The investigators will evaluate subject pre- and post training and at an interim point 3 weeks into the training sessions. The investigators anticipate that the VGRS will deliver more effective training by creating a realistic and challenging environment with accurate visual perception of a motor task which is being simultaneously performed by the user. The investigators will also gain an understanding of the rate of improvement for TT amputees during treadmill training. The research design will demonstrate the need for immersive virtual reality that includes a rich visual display and affords the opportunity to train on a variety of terrain conditions and mobility tasks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be unilateral transtibial amputees (TTA) between the ages of 18 and 65 who have consistently used a prosthesis for at least one year.
* Subjects must be community ambulators at a K3 level,

  * which dictates that they have the ability or potential to walk with variable cadence,
  * to traverse most environmental barriers and may have vocational, therapeutic, or exercise activity that demands prosthetic utilization beyond simple locomotion.

Exclusion Criteria:

* History of surgical procedures on their intact limb.
* Subjects will be excluded from the study if they present with

  * cardiovascular,
  * neurological,
  * or balance disorders that can affect gait.
  * Rheumatoid arthritis,
  * knee joint replacement,
  * and the use of ambulatory aids will also exclude participation.
* Subjects with considerable pain in their knee joints, as measured by a visual analog scale will also be excluded due to the confounding effects of pain on gait patterns.
* A medical history screening will be used to identify subjects with pre-existing conditions that would compromise their gait.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Knee Joint Symmetry at 6 weeks | Baseline and at 6 weeks
  Knee joint symmetry will be determined by joint loading (knee joint moments). Changes in joint loading will be measured as the difference in knee joint moment between the left and right leg (measured in Newtons/meter/kilogram of body weight).
Change from Baseline in Gait Speed (m/s) at 6 weeks | Baseline, at 3 weeks and at 6 weeks
  Gait speed (meters/second) will be measured while the participant is walking across a 40 foot walkway at a self selected speed
Change from Baseline in Gait Variability at 3 weeks and 6 weeks | Baseline, at 3 weeks and at 6 weeks
  Gait variability will be determined by calculating the magnitude of stride-to -stride fluctuations, normalized to each subject's mean stride time to define the Coefficient of Variation
Change from Baseline in Trunk Lean on the Prosthetic versus Non-Prosthetic Side of the Body (measured in degrees) at 6 weeks. | Baseline and at 6 weeks
  Gait symmetry will be determined by side to side trunk lean.

SECONDARY OUTCOMES:
Postural sway parameters - Swept Area - measured in meters x meters | Baseline and at 6 weeks
  To assess whole-body postural sway, displacement of the head-arm-trunk segment will be measured. The position of the center of mass (COM) of the body will be determined and the area swept by the COM will be calculated
Berg Balance Scale - clinical evaluation - scored on a scale of 0 -4 with a maximum score of 56 | Baseline and at 6 weeks
  The Berg Balance scale is used to measure balance by assessing the performance of functional tasks. Fourteen tasks are scored on a scale from 0 - 4 with 0 being less function and 4 reflecting the highest level of balance. Total score is 56.
  41-56 = low fall risk 21-40 = moderate fall risk 0 - 20 = high fall risk
Dynamic Gait Index - A four-point ordinal scale, ranging from 0-3 with a maximum score of 24. | Baseline and at 6 weeks
  Developed to assess the likelihood of a fall, the Dynamic Gait Index (DGI) is a four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. Eight different tasks are scored and the maximum score obtainable is 24 point.
  Interpretation: < 19/24 = predictive of falls; > 22/24 = safe ambulators
Four Square Step Test - the time it takes to step in four squares backwards, sideways and forward. Measured in seconds. | Baseline and at 6 weeks
  Test of dynamic balance that clinically assesses the person's ability to step over objects forward, sideways, and backwards
Postural sway parameters - Mediolateral excursion of the center of mass measured in millimeters | Baseline and at 6 weeks
  The maximum excursions and standard deviations of the center of mass trajectory in the Mediolateral direction of the body will be measured.
Postural sway parameters - Anteroposterior excursion of the center of mass measured in millimeters | Baseline and at 6 weeks
  The maximum excursions and standard deviations of the center of mass trajectory in the anteroposterior direction of the body will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E D'Andrea, PhD MS BS, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273